CLINICAL TRIAL: NCT04923503
Title: Department of Nutrition Science, Medical Faculty, Universitas Diponegoro, Semarang, Indonesia
Brief Title: Diurnal Ramadan Fasting on Appetite Hormone and Metabolic Profile Among Lean, Obesity, Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Etika Ratna Noer, Department of Nutrition, Medical Faculty, Universitas Diponegoro
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMD
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Fasting; Gut Hormone
Keywords: gut hormones; metabolic parameters; obesity; lean; diabetics; ramadan fasting
MeSH Terms: conditions — Fasting; Obesity

STUDY DESIGN:
Intervention Model Description: three arm parallel group with 45 subjects:
  1. fasting in lean group
  2. fasting in obese group
  3. fasting in diabetics group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: subject with random allocation Investigator do not know the group the analysator do not know the group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lean ramadan fasting (Experimental): conduct ramadan fasting for 30 days
  Interventions: Behavioral: diurnal fasting
- obese ramadan fasting (Experimental): conduct ramadan fasting for 30 days
  Interventions: Behavioral: diurnal fasting
- diabetics ramadan fasting (Experimental): conduct ramadan fasting for 30 days
  Interventions: Behavioral: diurnal fasting

INTERVENTIONS:
Behavioral: diurnal fasting — subject conduct fasting in Ramadan for 30 days
  Other Names: ramadan fasting

SUMMARY:
Diabetes Mellitus individuals are known to have dietary rules, namely regulating the amount, type and time of eating. Ramadan fasting seems to be beneficial for people who want to reduce their weight, but it is not easy for diabetic patients. Because of its distinctive features, Ramadhan induces changes in eating habits, calorie consumption, sleeping patterns, and daily physical activity, which may contribute to changes in hunger-satiety responses and glicemic control. Examining changes in gut hormones during Ramadan fasting may reveal whether this observance could change glucose metabolism in diabetics without triggering the undesirable effect of gluconeogenesis. The proportions of fat, protein, and carbohydrate in meals vary between outside and within Ramadan. Alterations in timing and composition meal during Ramadan lead to reduced food intake may affect gut hormones and metabolic responses. The aim of this study to determine whether the effect of Ramadan fasting differed in people with DM patients, pre-DM and healthy individuals, with respect to gut hormones, body composition, metabolic parameters, and glycemic control

DETAILED DESCRIPTION:
The experimental study was performed during and after Ramadan fasting in 2021 (April to May) in Semarang, Indonesia. The present study was performed using the quasy-experimental method by pre-post measurement of three experimental groups (diabetics, Obese and healthy subjects) selected using the purposive sampling methods

ELIGIBILITY:
Inclusion Criteria:

* Diabetics subjects: glucose fasting plasma > 200 mg/dL, with aged 35-60 years and body mass index above 25 kg/m;
* Obese subjects: body mass index above 25 kg/m2 with aged 35-60 years and waist circumference for men >90 cm, for women > 80 cm
* Lean subjects: body mass index below 23.5 kg/m2 with aged 35-60 years and waist circumference for men <90 cm, for women < 80 cm

Exclusion Criteria:

* experienced weight loss more than 10% from the actual weight in the last three months
* consumed medicine or supplement for weight loss diet, •. had the history of evidence of clinical depression, cognitive disorders, heart disease, cancer, liver or renal disease, chronic pulmonary disease, uncontrolled hypertension, physical disability, or other contraindications

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
change acylated ghrelin | 30 days
  Change from Baseline acyl ghrelin at 30 days taken in the lab from venous blood specimen
change PYY | 30 days
  Change from Baseline PYY at 30 days taken in the lab from venous blood specimen
change GLP-1 | 30 days
  Change from Baseline GLP-1 at 30 days taken in the lab from venous blood specimen
change insulin | 30 days
  Change from Baseline Insulin at 30 days taken in the lab from venous blood specimen

SECONDARY OUTCOMES:
change body weight | 30 days
  Change from Baseline body weight at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Etika R Noer, Principal Investigator — Diponegoro University
Locations (1):
- Etika Ratna Noer, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the result of this study is available to cite everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: anytime
Access Criteria: etikaratna@fk.undip.ac.id
URL: http://dept-gizi@fk.undip.ac.id